CLINICAL TRIAL: NCT05934461
Title: A Retrospective Study of Radiotherapy Combined With EGFR-TKI for Stage III EGFR Mutant Lung Cancer
Status: Completed | Type: Observational
Sponsor: Laibin People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Gang, Deputy Director of the Department of Oncology, Laibin People's Hospital
Other Study IDs: Z-G20221781
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-12

CONDITIONS: The Primary Study Metric is Progression-free Survival (PFS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- an open-label, multiinstitutional, single-arm retrospective study: Three-dimensional conformal radiotherapy (3DCRT) or intensity-modulated conformal radiotherapy (IMRT) at a prescribed dose of 54-66 Gy/27-33 f. The combined TKI includes gefitinib, erlotinib, erlotinib, oseltinib, and ametinib. The specific uses are: gefitinib 250 mg orally once daily; erlotinib 125 mg orally three times daily; erlotinib 150 mg orally once daily; oseltinib 80 mg orally once daily; ametinib 110 mg orally once daily. TKI is taken until disease progression or intolerability.
- RT+C: Three-dimensional conformal radiotherapy (3DCRT) or intensity-modulated conformal radiotherapy (IMRT) at a prescribed dose of 54-66 Gy/27-33 f. The combined TKI includes gefitinib, erlotinib, erlotinib, oseltinib, and ametinib. The specific uses are: gefitinib 250 mg orally once daily; erlotinib 125 mg orally three times daily; erlotinib 150 mg orally once daily; oseltinib 80 mg orally once daily; ametinib 110 mg orally once daily. TKI is taken until disease progression or intolerability.

SUMMARY:
Objective: To investigate the efficacy and safety of radiotherapy combined with EGFR-KI in the treatment of stage III EGFR mutant lung cancer. Methods: Stage III EGFR mutant lung cancer cases who underwent radiotherapy combined with EGFR-TKI from December 2014 to December 2022 at the People's Hospital of Laibin, the First People's Hospital of Yulin, the Affiliated Hospital of Guilin Medical College, and the Park East Hospital of Guangxi Medical University Kaiyuan were collected, and the primary index of the study was progression-free survival (PFS), and the secondary indexes were objective remission rate, overall survival, recurrence pattern, and adverse events. Survival analysis was performed using the Kaplan-Meier method with Log rank test for univariate analysis and Cox proportional risk model for multifactorial analysis of prognosis.

ELIGIBILITY:
Inclusion Criteria:

* ①patients diagnosed with lung cancer by pathology; ②genetic testing for EGFR mutation type; ③compliance with the international eighth edition of lung cancer TNM stage IIIA-IIIC; ④treatment modality of radiotherapy + targeted therapy. ⑤Eastern Cooperative Oncology Group (ECOG) physical status score ≤ 2

Exclusion Criteria:

* (1) those who underwent surgery; (2) those who received chemotherapy. (3) Combination of other serious diseases that affect survival.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with lung cancer by pathology,genetic testing for EGFR mutation type
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 years
  the time from treatment initiation to first documented progressive disease (PD) or time to death.